CLINICAL TRIAL: NCT06486246
Title: Geniculate Nerve Block Versus Adductor Canal Block for ACL Reconstruction Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Xavier Sala-Blanch, Principal investigator, Hospital Clinic of Barcelona
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LCAGEN1
Record Dates: First submitted 2024-05-02; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: ACL Tear; Pain, Postoperative
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: UNIcenter Non-randomized trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adductor canal block (Experimental): Injection of local anaesthetics under ultrasound guidance in the adductor canal by the anaesthesiologist prior the surgery, after inducction of general anesthesia.
  Interventions: Procedure: Adductor canal block
- Genicular nerve block (Experimental): Injection of local anaesthetics under ultrasound guidance in the genicular nerves ( Superomedial genicular nerve, superolateral genicular nerve and inferomedial genicular nerve) by the anaesthesiologist prior the surgery, after inducction of general anesthesia.
  Interventions: Procedure: Adductor canal block

INTERVENTIONS:
Procedure: Adductor canal block — Injection of the local anesthetic prior to the surgery, either in the the adductor canal or in the genicular nerves by the anesthesiologist under ultrasound guidance.
  Other Names: Genicular nerve block

SUMMARY:
Anterior cruciate ligament repair (ACL) surgery presents moderate to severe pain during the inmediate postoperative period and the first days after surgery. In addition, due to the interest of surgeons and patients for early reinstatement, the use of blockages that decrease the strength of the quadriceps is avoided. Therefore, in recent years, the adductor canal block (ACB) has been used for postoperative analgesia with variable results.

Genicular nerve block (GNB) has been used for pain management in patients with knee osteoarthritis and recently in knee arthroplasty surgery with results similar to the local anesthetic infiltration techniques by the surgeon (LIA). Considering their good results in these patients in addition to being a 100% sensitive block without risk of motor involvement.

The investigators proposed this experimental study to evaluate tha analgesic efficacy of the genicular nerve block (GNB) compared with the adductor canal block (ACB) for the Anterior cruciate ligament (ACL) repair surgery.

DETAILED DESCRIPTION:
Participants scheduled to undergo anterior cruciate ligament reconstruction under general anaesthesia will be allocated to two groups: Adductor canal block or Genicular nerve block- The adductor canal block will be performed by the anaesthesiologist under ultrasound guidance prior the surgery, after inducction , using 20 mLs Ropivacaine 0.2%. The genicular nerve block will be performed by the anaesthesiologist under ultrasound guidance prior the surgery, after inducction , using 20 mLs Ropivacaine 0.2% in total.

Postoperative analgesia will include analgesia (Dexketoprofen 75 mg during first 24 hours), acetomiophen 1 gr every 8 hours and tramadol for rescue pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 18 to 50 years old scheduled to undergo anterior cruciate ligament reconstruction

Exclusion Criteria:

* peripheral neuropathy
* pre-existing femoral neuropathy
* diabetes mellitus
* alcoholism
* drug addiction
* cancer with chemotherapy
* chronic pain state
* Negative of the patient to participate in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain assessed by NRS at PACU | up to 6 hours postoperative
  Numerical raiting score (NRS) 0-10 (0= No pain; 10=maximum pain)
Opioid consumption at PACU | up to 6 hours postoperative
  Metadone consumption in mg.

SECONDARY OUTCOMES:
Pain score at home | up to 24 hours
  Numerical raiting score (NRS) 0-10 (0= No pain; 10=maximum pain)
Quality of rest | First night
  Sleep or wake-up during first night (Pain) (Awake because of pain: Yes / NO)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic, Barcelona, Spain